CLINICAL TRIAL: NCT00555256
Title: A Phase I Study of SUNITINIB and Rapamycin in Advanced Non-Small Cell Lung Cancer (NSCLC)
Acronym: SU/Rapamycin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-0562 / 201101709
Record Dates: First submitted 2007-11-07; First posted 2007-11-08 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2013-03

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Sunitinib; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Patients will be instructed to take sunitinib and rapamycin every morning for 4 weeks, then to take 2 weeks off. The sunitinib dose will be 25mg in the first cohort and the rapamycin dose will be 2 mg.
  Interventions: Drug: sunitinib and rapamycin (Drug will be held)

INTERVENTIONS:
Drug: sunitinib and rapamycin (Drug will be held) — Any toxicity causing a total of 14 days delay of therapy will be considered dose limiting.

SUMMARY:
To define the optimal dose of sunitinib when given in combination with rapamycin 2mg.

To determine the maximum tolerated dosage of sunitinib and rapamycin given in this fashion.

To determine the how many times and how severe other toxicities of this combination therapy.

To determine how quickly the patient(s) will respond the the drug, overall survival and time to progression for this combination therapy.

DETAILED DESCRIPTION:
We propose to conduct a phase I study of sunitinib and rapamycin administered daily for weeks 1-4)in a 6-week cycle. The rationale for this study includes:

* Sunitinib is a tyrosine kinase inhibitor that targets multiple receptor pathways critical for cell growth. It has both antiangiogenic and direct antitumor activities.
* Resistance to receptor tyrosine kinase inhibitors is well-documented. The mammalian target of rapamycin (mTOR) pathway may play a critical role in imatinib-refractory GIST. Rapamycin and other agents that inhibit mTOR demonstrate antiangiogenic and antitumor properties by decreasing VEGF production and decreasing responsiveness to VEGF.
* Sunitinib is approved and well-tolerated at doses as high as 75mg daily. The typical dose in most Phase II and III trials has been 50mg/day, given on a four weeks on/two weeks off schedule. There are, however, recent trials looking at a lower dosage, 37.5 mg, in NSCLC.
* Rapamycin at doses greater than 2 mg daily is documented to be well-tolerated in renal transplant patients. In renal transplant patients, 2mg daily is the typical starting dose. This dose was used in one of the phase I studies of rapamycin in glioblastoma.
* The administration of two oral medications, taken once daily, may be more convenient to patients than iv administration of chemotherapy at an infusion center every 1-3 weeks.
* Based on these data, initial dosing of sunitinib beginning at 37.5 mg orally everyday for 4 weeks, followed by 2 weeks off, in combination with rapamycin 2 mg/day orally for 6 weeks during a 6 week cycle should be well tolerated and allow for dose-finding escalation.

ELIGIBILITY:
* Patients must have a histologically or cytologically proven NSCLC, including adenocarcinoma, broncho-alveolar cell and large cell anaplastic carcinoma
* Patients need not have measurable disease to be eligible for this study. Patients with non-measurable lesions will be eligible. Measurable and non-measurable disease will be defined by RECIST criteria
* Age ≥18 years
* ECOG 0-2
* Life Expectancy: ≥3 months
* Patients who have had prior therapy must have completed chemotherapy at least 3 weeks, and radiotherapy at least 2 weeks, prior to study drug administration, with all side effects resolved. Patients who have not received prior therapy are eligible if they are not good candidates for standard treatment with cytotoxic chemotherapy, or do not wish to receive cytotoxic chemotherapy.
* Patients may not have undergone major surgery within 4 weeks prior to starting study drug administration. In addition, any surgical complications must be resolved, and the surgical scar must be determined by the surgeon to be healing appropriately
* Patients must have recovered from uncontrolled intercurrent illness including, but not limited to, ongoing active infection
* Patients may not have had any of the following within 6 months prior to study drug administration: MI, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic CHF, CVA, TIA or PE
* Patients may not have had a grade 3 hemorrhage within 4 weeks of study drug administration
* Patients may not have a history of or active spinal cord compression or carcinomatous meningitis. In addition, any previous brain metastases should be adequately treated, and there should be no evidence of new brain or leptomeningeal metastases on a screening CT or MRI scan
* Patients may not have ongoing cardiac dysrhythmias of grade ≥2. In addition, they may not have a prolonged QTc interval on baseline EKG
* Patients may not have uncontrolled hypertension or thyroid disease
* Patients may not have a severe acute or chronic medical or psychiatric condition, or laboratory abnormality
* Patients must have adequate bone marrow function defined as an absolute neutrophil count ≥ 1,500 cells/mm3, Hgb ≥ 9g/dl and platelet count ≥ 100,000 cells/mm3
* Patients must have adequate liver function defined as bilirubin <=2 x the upper limit of institutional normal and SGOT and SGPT <=2.5 x the upper limit of institutional normal, or SGOT and SGPT <=5 x the upper limit of institutional normal if liver function abnormalities are due to underlying malignancy
* Patients must have adequate renal function defined as serum creatinine <=1.5 x the upper limit of institutional normal
* Patients must have serum calcium ≤12.0 mg/dL
* No previous history of severe hypersensitivity reaction attributed to a receptor tyrosine kinase inhibitor.
* For all patients with reproductive potential, the use of adequate contraception and will be required for the duration of treatment and the 3 months following treatment
* Pregnant and nursing women are not eligible
* After being informed of the treatment involved, patients must give written consent. The patient should not have any serious medical or psychiatric illness that would prevent either the giving of informed consent or the receipt of treatment
* Entry to this study is open to both men and women and to all racial and ethnic subgroups

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-11; Primary Completion 2010-02 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To define the optimal dose of sunitinib when given in combination with rapamycin 2mg daily. | 6 weeks
Determine the dose limiting toxicity of sunitinib and rapamycin | 6 weeks

SECONDARY OUTCOMES:
Incidence and severity of other toxicities | 30 days after the end of treatment
  Cycles are 6 weeks long and can have as many as 9 cycles
Response rates | 30 days after end of treatment
Overall survival | 12 months from date of first treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ramaswamy Govindan, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Jemal A, Murray T, Ward E, Samuels A, Tiwari RC, Ghafoor A, Feuer EJ, Thun MJ. Cancer statistics, 2005. CA Cancer J Clin. 2005 Jan-Feb;55(1):10-30. doi: 10.3322/canjclin.55.1.10. PMID 15661684
- [Background] Shepherd FA, Rodrigues Pereira J, Ciuleanu T, Tan EH, Hirsh V, Thongprasert S, Campos D, Maoleekoonpiroj S, Smylie M, Martins R, van Kooten M, Dediu M, Findlay B, Tu D, Johnston D, Bezjak A, Clark G, Santabarbara P, Seymour L; National Cancer Institute of Canada Clinical Trials Group. Erlotinib in previously treated non-small-cell lung cancer. N Engl J Med. 2005 Jul 14;353(2):123-32. doi: 10.1056/NEJMoa050753. PMID 16014882
- [Background] Abrams TJ, Lee LB, Murray LJ, Pryer NK, Cherrington JM. SU11248 inhibits KIT and platelet-derived growth factor receptor beta in preclinical models of human small cell lung cancer. Mol Cancer Ther. 2003 May;2(5):471-8. PMID 12748309
- [Background] O'Farrell AM, Abrams TJ, Yuen HA, Ngai TJ, Louie SG, Yee KW, Wong LM, Hong W, Lee LB, Town A, Smolich BD, Manning WC, Murray LJ, Heinrich MC, Cherrington JM. SU11248 is a novel FLT3 tyrosine kinase inhibitor with potent activity in vitro and in vivo. Blood. 2003 May 1;101(9):3597-605. doi: 10.1182/blood-2002-07-2307. Epub 2003 Jan 16. PMID 12531805
- [Background] McKeage MJ, Raynaud F, Ward J, Berry C, O'Dell D, Kelland LR, Murrer B, Santabarabara P, Harrap KR, Judson IR. Phase I and pharmacokinetic study of an oral platinum complex given daily for 5 days in patients with cancer. J Clin Oncol. 1997 Jul;15(7):2691-700. doi: 10.1200/JCO.1997.15.7.2691. PMID 9215842
- [Background] Heinrich MC, Corless CL, Demetri GD, Blanke CD, von Mehren M, Joensuu H, McGreevey LS, Chen CJ, Van den Abbeele AD, Druker BJ, Kiese B, Eisenberg B, Roberts PJ, Singer S, Fletcher CD, Silberman S, Dimitrijevic S, Fletcher JA. Kinase mutations and imatinib response in patients with metastatic gastrointestinal stromal tumor. J Clin Oncol. 2003 Dec 1;21(23):4342-9. doi: 10.1200/JCO.2003.04.190. PMID 14645423
- [Background] Kulke, M., et al., A phase 2 study to evaluate the efficacy and safety of SU11248 in patients (pts) with unresectable neuroendocrine tumors (NETs). J Clin Oncol (Meeting Abstracts), 2005. 23(16_suppl): p. 4008-.
- [Background] Lenz, H., et al., Phase II trial of SU11248 in patients with metastatic colorectal cancer (MCRC) after failure of standard chemotherapy. ASCO Gastrointestinal Cancers Symposium, 2006: p. Abst. No. 241.
- [Background] Motzer RJ, Michaelson MD, Redman BG, Hudes GR, Wilding G, Figlin RA, Ginsberg MS, Kim ST, Baum CM, DePrimo SE, Li JZ, Bello CL, Theuer CP, George DJ, Rini BI. Activity of SU11248, a multitargeted inhibitor of vascular endothelial growth factor receptor and platelet-derived growth factor receptor, in patients with metastatic renal cell carcinoma. J Clin Oncol. 2006 Jan 1;24(1):16-24. doi: 10.1200/JCO.2005.02.2574. Epub 2005 Dec 5. PMID 16330672
- [Background] Socinski, M.A., et al., Efficacy and safety of Sunitinib in previously treated, advanced non-small cell lung cancer (NSCLC): Preliminary results of a multicenter, phase II trial. Proc Am Soc Clin Oncol, 2006: p. Abst. 7001.
- [Background] Casali, P.G., et al. Updated results from a phase III trial of Sunitinib in GIST patients (pts) for whom imatinib (IM) therapy has failed due to resistance or intolerance. in Proc Am Soc Clin Oncol. 2006.
- [Background] Motzer, R.J., et al., Phase III randomized trial of Sunitinib (SU11248) versus interferon-alfa (IFN-a) as first-line systemic therapy for patients with metastatic renal cell carcinoma (mRCC). Proc Am Soc Clin Oncol, 2006: p. Abst. LBA3.
- [Background] Guba M, von Breitenbuch P, Steinbauer M, Koehl G, Flegel S, Hornung M, Bruns CJ, Zuelke C, Farkas S, Anthuber M, Jauch KW, Geissler EK. Rapamycin inhibits primary and metastatic tumor growth by antiangiogenesis: involvement of vascular endothelial growth factor. Nat Med. 2002 Feb;8(2):128-35. doi: 10.1038/nm0202-128. PMID 11821896
- [Background] Smolewski P. Recent developments in targeting the mammalian target of rapamycin (mTOR) kinase pathway. Anticancer Drugs. 2006 Jun;17(5):487-94. doi: 10.1097/00001813-200606000-00001. PMID 16702804
- [Background] Busca R, Bertolotto C, Ortonne JP, Ballotti R. Inhibition of the phosphatidylinositol 3-kinase/p70(S6)-kinase pathway induces B16 melanoma cell differentiation. J Biol Chem. 1996 Dec 13;271(50):31824-30. doi: 10.1074/jbc.271.50.31824. PMID 8943224
- [Background] Mayerhofer M, Aichberger KJ, Florian S, Krauth MT, Hauswirth AW, Derdak S, Sperr WR, Esterbauer H, Wagner O, Marosi C, Pickl WF, Deininger M, Weisberg E, Druker BJ, Griffin JD, Sillaber C, Valent P. Identification of mTOR as a novel bifunctional target in chronic myeloid leukemia: dissection of growth-inhibitory and VEGF-suppressive effects of rapamycin in leukemic cells. FASEB J. 2005 Jun;19(8):960-2. doi: 10.1096/fj.04-1973fje. Epub 2005 Mar 22. PMID 15784722
- [Background] Grewe M, Gansauge F, Schmid RM, Adler G, Seufferlein T. Regulation of cell growth and cyclin D1 expression by the constitutively active FRAP-p70s6K pathway in human pancreatic cancer cells. Cancer Res. 1999 Aug 1;59(15):3581-7. PMID 10446965
- [Background] Shapira M, Kakiashvili E, Rosenberg T, Hershko DD. The mTOR inhibitor rapamycin down-regulates the expression of the ubiquitin ligase subunit Skp2 in breast cancer cells. Breast Cancer Res. 2006;8(4):R46. doi: 10.1186/bcr1533. PMID 16859513
- [Background] Chang SM, Wen P, Cloughesy T, Greenberg H, Schiff D, Conrad C, Fink K, Robins HI, De Angelis L, Raizer J, Hess K, Aldape K, Lamborn KR, Kuhn J, Dancey J, Prados MD; North American Brain Tumor Consortium and the National Cancer Institute. Phase II study of CCI-779 in patients with recurrent glioblastoma multiforme. Invest New Drugs. 2005 Aug;23(4):357-61. doi: 10.1007/s10637-005-1444-0. PMID 16012795
- [Background] Margolin K, Longmate J, Baratta T, Synold T, Christensen S, Weber J, Gajewski T, Quirt I, Doroshow JH. CCI-779 in metastatic melanoma: a phase II trial of the California Cancer Consortium. Cancer. 2005 Sep 1;104(5):1045-8. doi: 10.1002/cncr.21265. PMID 16007689
- [Background] Galanis E, Buckner JC, Maurer MJ, Kreisberg JI, Ballman K, Boni J, Peralba JM, Jenkins RB, Dakhil SR, Morton RF, Jaeckle KA, Scheithauer BW, Dancey J, Hidalgo M, Walsh DJ; North Central Cancer Treatment Group. Phase II trial of temsirolimus (CCI-779) in recurrent glioblastoma multiforme: a North Central Cancer Treatment Group Study. J Clin Oncol. 2005 Aug 10;23(23):5294-304. doi: 10.1200/JCO.2005.23.622. Epub 2005 Jul 5. PMID 15998902
- [Background] Chan S, Scheulen ME, Johnston S, Mross K, Cardoso F, Dittrich C, Eiermann W, Hess D, Morant R, Semiglazov V, Borner M, Salzberg M, Ostapenko V, Illiger HJ, Behringer D, Bardy-Bouxin N, Boni J, Kong S, Cincotta M, Moore L. Phase II study of temsirolimus (CCI-779), a novel inhibitor of mTOR, in heavily pretreated patients with locally advanced or metastatic breast cancer. J Clin Oncol. 2005 Aug 10;23(23):5314-22. doi: 10.1200/JCO.2005.66.130. Epub 2005 Jun 13. PMID 15955899
- [Background] Atkins MB, Hidalgo M, Stadler WM, Logan TF, Dutcher JP, Hudes GR, Park Y, Liou SH, Marshall B, Boni JP, Dukart G, Sherman ML. Randomized phase II study of multiple dose levels of CCI-779, a novel mammalian target of rapamycin kinase inhibitor, in patients with advanced refractory renal cell carcinoma. J Clin Oncol. 2004 Mar 1;22(5):909-18. doi: 10.1200/JCO.2004.08.185. PMID 14990647
- [Background] Okuno, S.H., et al., A multicenter phase consortium (P2C) study of the mTOR inhibitor CCI-779 in advanced soft tissue sarcomas (STS). Proc Am Soc Clin Oncol, 2006.
- [Background] Pandya, K.J., et al., A randomized, phase II ECOG trial of two dose levels of temsirolimus (CCI-779) in patients with extensive stage small cell lung cancer in remission after induction chemotherapy. A preliminary report. ASCO Proceedings, 2005: p. Abstract No: 7005.
- [Background] MacDonald AS. Rapamycin in combination with cyclosporine or tacrolimus in liver, pancreas, and kidney transplantation. Transplant Proc. 2003 May;35(3 Suppl):201S-208S. doi: 10.1016/s0041-1345(03)00231-8. PMID 12742497
- [Background] Reardon DA, Quinn JA, Vredenburgh JJ, Gururangan S, Friedman AH, Desjardins A, Sathornsumetee S, Herndon JE 2nd, Dowell JM, McLendon RE, Provenzale JM, Sampson JH, Smith RP, Swaisland AJ, Ochs JS, Lyons P, Tourt-Uhlig S, Bigner DD, Friedman HS, Rich JN. Phase 1 trial of gefitinib plus sirolimus in adults with recurrent malignant glioma. Clin Cancer Res. 2006 Feb 1;12(3 Pt 1):860-8. doi: 10.1158/1078-0432.CCR-05-2215. PMID 16467100
- [Background] Das, A., et al., Phase I study of Gefitinib and rapamycin in patients with recurrent or progressive glioblastoma (GBM). ASCO Proceedings, 2005.
- [Result] Fletcher, J.A., et al., Mechanisms of resistance to imatinib mesylate (IM) in advanced gastrointestinal stromal tumor (GIST). Proc Am Soc Clin Oncol, 2003. 22: p. page 815, (abstr 3275).
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu